CLINICAL TRIAL: NCT05555225
Title: Methylome Study in Patients Affected With Sporadic Limb Malformations
Brief Title: Methylome Study in Sporadic Limb Malformations
Acronym: METHYLIMB
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0524; 2022-A01441-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-09-23; First posted 2022-09-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Amelia; Femur Fibula Ulna Syndrome
Keywords: Amelia; Femur-Fibula-Ulna Syndrome; Methylation; Limb development; Gene regulation
MeSH Terms: conditions — Ectromelia; Femur fibula ulna syndrome | interventions — Epigenome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with amelia: Patients with severe hypoplasia or agenesia of at least two limbs who gave their consent for the research and for whom a DNA sample is available in our laboratory
  Interventions: Other: Methylome
- Patients with Femur-Fibula-Ulna Syndrome: Patients with anomaly of at least one femur, one fibula and with oligodactyly who gave their consent for the research and for whom a DNA sample is available in our laboratory.
  Interventions: Other: Methylome
- Healthy subjects: Healthy subjects used as controls, who gave their consent for the research and for whom a DNA sample is available in our laboratory.
  Interventions: Other: Methylome

INTERVENTIONS:
Other: Methylome — Epigenetic study : analysis of DNA methylation

SUMMARY:
Some limb malformations are known to be sporadic (non hereditary). For these malformations, no molecular cause was identified, even after whole genome sequencing. Methylation of CpG islands is an epigenetic process which is usually not transmitted to the descents. We hypothesize that sporadic limb malformations may be due to a methylation anomaly. This study will include patients with Amelia or Femur Fibula Ulna Syndrome. With patients consent, we will study the methylome on DNA samples already available in our laboratory. Each patient sample will be paired to a control of same tissue, age and sex. By bioinformatics comparison, we will identify differentially methylated candidate regions.

ELIGIBILITY:
Inclusion Criteria:

* Specific consent for this study
* DNA available in the laboratory
* For amelia : agenesia of 2 or 4 limbs
* For Femur-Fibula-Ulna Syndrome : hypoplasia or agenesia of the femur uni or bilateral with hypoplasia or agenesia or bowing of the fibula and/or of the ulna

Exclusion Criteria:

* No consent
* No available DNA or poor quality of the DNA sample
* Patient under tutorship
* Pregnancy or nursing mother
* Patient non covered by the French social security

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: DNA samples were obtained from the molecular biology laboratory of Lille university hospital. All patients exhibiting amelia or Femur-Fibula-Ulna Syndrome and with enough DNA available in the lab could be included.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Differentially Methylated Regions | through study completion an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Perrine BRUNELLE, MD, Principal Investigator — University Hospital, Lille